CLINICAL TRIAL: NCT07218211
Title: INCLUSION - Enhancing PrEP Uptake and Retention Among Latine Transgender Women and Gay, Bisexual, and Other Men Who Have Sex With Men in the South Using Long-Acting Injectable PrEP
Brief Title: Enhancing PrEP Uptake and Retention Among Latine TGW and GBM in the South Using Long-Acting Injectable PrEP
Acronym: INCLUSION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00118575
Record Dates: First submitted 2025-10-03; First posted 2025-10-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: HIV Prevention; HIV Pre-exposure Prophylaxis; HIV Prevention Program; HIV Prevention and Care; HIV Pre-exposure Prophylaxis Use
Keywords: Long-acting Injectable PrEP; Lenacapavir; PrEP; PrEP injections
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long-acting Injectable PrEP (lenacapavir) program (Other): Community-delivered long-acting injectable PrEP (lenacapavir) program for Latine gay and bisexual men (GBM) and transgender women (TGW)
  Interventions: Drug: Lenacapavir long-acting

INTERVENTIONS:
Drug: Lenacapavir long-acting — Culturally-tailored, community-delivered long-acting injectable PrEP (lenacapavir)
  Other Names: Yeztugo; Lenacapavir injection; PrEP; Injectable PrEP

SUMMARY:
The purpose of this project is to test a culturally-tailored, community-delivered long-acting injectable PrEP (lenacapavir) program for Latine gay and bisexual men (GBM) and transgender women (TGW). The objective is to evaluate whether this intervention demonstrates greater persistence on lenacapavir for Latine GBM and TGW compared with what has been observed historically at the Duke PrEP Clinic.

DETAILED DESCRIPTION:
We propose a mixed methods hybrid type 3 implementation study, which primarily tests an implementation strategy while collecting data on the clinical intervention and related outcomes. Building on existing partnerships between Duke University and El Centro Hispano, we will integrate lenacapavir delivery on-site at El Centro Hispano facilities, leveraging El Centro Hispano Peer Navigators to provide culturally congruent support for PrEP uptake, adherence, and persistence among Latine GBM and TGW.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be assigned male sex at birth.
* Report sexual activity with a someone assigned male at birth OR identify as GBM or TGW; be HIV-negative.
* Identify as Hispanic and/or Latine .
* Be able to provide informed consent in English or Spanish .
* Be 18 years or older .
* Weigh at least 77 lbs (35 kg) by self-reported weight.
* Interested in PrEP and willing to undergo the study procedures.

Exclusion Criteria:

* Individuals living with HIV.
* Individuals assigned female sex at birth will be excluded.
* Individuals who are currently taking oral PrEP from another source and are not willing to switch to lenacapavir for PrEP for the duration of the study will also be excluded.
* Individuals who report a history of severe renal or hepatic disease or with clinical stigmata of either disease on physical exam as assessed by a study clinician will be excluded.
* Individuals taking a medication with a significant interaction with lenacapavir will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Latine gay and bisexual men (GBM) and transgender women (TGW)
Enrollment: 100 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who provided identification of barriers to providing lenacapavir at a Latine community-based organization | up to 1 year
  Qualitative identification: "What gets in the way of people in your community starting PrEP? Staying on PrEP?"
Number of participants who provided recommendations to address barriers to providing lenacapavir at a Latine community-based organization | up to 1 year
  Qualitative identification: "Recommendations to address these barriers?"
Number of participants who provided identification of facilitators to providing lenacapavir at a Latine community-based organization | up to 1 year
  Qualitative identification: "What factors support people in your community?"

SECONDARY OUTCOMES:
Acceptability as measured by the number of participants who answered "yes" to select modified acceptability questions from Abbreviated Acceptability Rating Profile (AARP) | up to 1 year
  AARP items will help quantify acceptability and will help validate community perceptions: "I believe lenacapavir injections are an effective way to prevent HIV", "I would be willing to receive lenacapavir injections in the future when this study is complete", "Receiving lenacapavir in a community setting fits my lifestyle and preferences", "I feel comfortable receiving lenacapavir injections from professionals working with El Centro", "I would recommend lenacapavir to a friend who is at risk for HIV", "I found lenacapavir preferable to oral PrEP", "Compared to a daily pill, I feel that injectable PrEP gives me more privacy", "I am concerned about possible side effects from lenacapavir injections", "Compared to a daily pill, I feel that injectable PrEP reduces concerns about being judged by others"
Number of providers who found the intervention feasible as measured by the Program Sustainability Assessment Tool (PSAT) | up to 1 year
  The PSAT will provide a structured way to assess organizational capacity and sustainability for scale up. It has a score range of 0 to 40, where a higher score indicates greater feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Tonia Poteat, PhD, Principal Investigator — Duke University Medical Center - Professor in the School of Nursing
Locations (1):
- El Centro Hispano, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No